CLINICAL TRIAL: NCT01365702
Title: Clinical Efficacy of Tiotripium in Patients With Airflow Obstruction Due to TB Destroyed Lung
Brief Title: Tiotropium in Patients With Tuberculosis (TB) Destroyed Lung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sei Won Lee/Assistant professor, Department of Internal Medicine, Seoul National University Bundang Hospital
Other Study IDs: SNUBH_TLD and spiriva
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Lung Disease, Obstructive; Tuberculosis
Keywords: COPD; tiotropium; tuberculous destroyed lung
MeSH Terms: conditions — Lung Diseases, Obstructive; Tuberculosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tiotropium in TB destroyed lung

SUMMARY:
The aim of this study to evaluate clinical efficacy of tiotropium in patients with airflow obstruction due to Tuberculosis (TB) destroyed lung.

DETAILED DESCRIPTION:
Tuberculosis can cause lung parenchymal destruction, volume loss, secondary bronchiectasis. Patients with TB destroyed lung complain chronic respiratory symptoms, such as chronic cough, sputum, dyspnea, exercise intolerance, and acute exacerbations. Some of them have chronic airflow obstructions on pulmonary function tests, similar to those of smokers.

Previous large randomized controlled trials, targeting patients with smoking related moderate to severe COPD,demonstrated that tiotropium improved quality of life and respiratory symptom with tolerable long-term safety. The investigators want to evaluate whether tiotropium can improve chronic respiratory symptom,an lung function in patients with COPD due to TB destroyed lung.

ELIGIBILITY:
Inclusion Criteria:

* previous pulmonary tuberculosis history
* never smoker or light smoker (<10 pack-year)
* destruction of lung parenchyme, lung volume loss,secondary bronchiectasis due to tuberculosis in chest radiographs or chest CT, confirmed by board-certificate radiologist
* airflow obstruction confirmed by pulmonary function test, FEV1/FVC <70%

Exclusion Criteria:

* patients do not agree with study enrollment
* patients with active tuberculosis or current antituberculous medication
* patients under chemotherapy or other immunosuppressant therapy such as glucocorticoid.
* active infection such as pneumonia, tuberculosis
* patients who are illiterate
* patients with dementia
* pregnant or to be pregnant
* previous lung resection surgery history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with TB destroyed lung visiting Seoul National University Bundang Hospital Respiratory center for chronic respiratory symptoms will be screened for study participants. Among the patients, those with definite pulmonary TB histor with airflow obstruction on their PFT were entrolled.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
St-George respiratory questionnaire(SGRQ) | 6 months after initiation of tiotropium once-daily inhalation

SECONDARY OUTCOMES:
lung function | 6mo after initiation of tiotropium once-daily inhalation
cough VAS | 6mo after initiation of tiotropium once-daily inhalation
adverse reaction of tiotropium | 6 months after initiation of tiotropium once-daily inhalation

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, M.D., Principal Investigator — Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical research center, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea